CLINICAL TRIAL: NCT06555211
Title: Cardio and Renovascular Effects of Static Muscle Work in the Healthy Human - Measured With Finapres® and Positron Emission Tomography (PET) Using 15-oxygen Labeled Water as Tracer Compared to Magnetic Resonance (MR)
Brief Title: Cardio and Renovascular Effects of Isometric Exercise in the Healthy Human Measured by PET/CT and MRI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bispebjerg Hospital (Other)
Responsible Party: Principal Investigator, Ali Asmar, Chief Physician, Associate Professor, Bispebjerg Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: H-23037460
Record Dates: First submitted 2024-08-07; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Kidneys
Keywords: Total renal blood flow; Regional renal perfusion; Regional renal oxygenation; Renal oxygen extraction

STUDY DESIGN:
Intervention Model Description: Each participant will undergo intervention, which is PET/CT, and control, which is MRI. Each participant will have both intervention and control performed the same day in randomized order.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group randomized to begin with MRI (Other): Group is randomized to begin with MRI and have PET/CT performed later on the same day
  Interventions: Procedure: MRI; Procedure: PET/CT
- Group randomized to begin with PET/CT (Other): Group is randomized to begin with PET/CT and have MRI performed later on the same day
  Interventions: Procedure: MRI; Procedure: PET/CT

INTERVENTIONS:
Procedure: MRI — MRI will be performed
Procedure: PET/CT — PET/CT will be performed

SUMMARY:
This randomized crossover study aims to validate measurements of renal perfusion in healthy males with PET/CT, using 15-oxygen labeled water as tracer, against the validated multiparametric MRI technique.

The study will determine:

* Total renal blood flow and regional renal perfusion at baseline (rest) and during isometric muscle exercise of the upper arm, using PET/CT (with 15-oxygen labeled water as a tracer) and MRI.
* The coefficient of variation of renal blood flow and regional renal perfusion measurements at baseline and during isometric muscle exercise of the upper arm, using PET/CT (with 15-oxygen labeled water as a tracer) and MRI.
* Regional renal oxygenation and oxygen extraction at baseline and during isometric muscle exercise of the upper arm using MRI.
* The coefficient of variation on regional renal oxygenation and oxygen extraction measurements at baseline and during isometric muscle exercise of the upper arm using MRI.

DETAILED DESCRIPTION:
Measuring tissue perfusion with PET/CT using 15-oxygen labeled water is routinely used as a non-invasive tool to examine cerebral and myocardial perfusion. With a 100% tissue extraction, 15-oxygen labeled water is gold standard.

The aim of the present study is to validate renal perfusion measurements with PET/CT using 15-oxygen labeled water as tracer against the validated multiparametric MRI technique.

Once validated the imaging technique will be beneficial in examining vascular damage in the kidneys caused by different renal diseases.

This is a randomized, crossover study where each participant will participate in 1 study day.

Ten healthy male participants in the age group 20-60 years are screened and randomized, and expected to complete the present study. Informed consent is obtained before the screening meeting.

All participants consume a controlled diet with fixed salt intake corresponding to a daily intake of 50-70 mmol + 2 mmol/kg sodium for 4 days before the experiment. On the fourth day, 24-hour urine collection will be performed. Throughout the 4 day period, water intake will be ad libitum and physical activity will not be allowed.

Each participant will undergo both PET/CT and MRI separated by around 1.5 hour.

Total renal blood flow and regional renal perfusion are measured repeatedly altogether 5 times with both PET/CT and MRI. Renal oxygenation and oxygen extraction are measured repeatedly 5 times as well, using MRI. The 5 measurements consist of 2 at baseline (rest), 2 during isometric exercise (handgrip) and 1 during recovery (rest).

Isometric muscle exercise is conducted by squeezing a handgrip coupled to a dynamometer. This increases sympathetic nervous activity, leading to preglomerular vasoconstriction.

ELIGIBILITY:
Inclusion Criteria:

* Normal health stated through medical questionnaire, examination and blood samples.

Exclusion Criteria:

* Immunosuppressive treatment
* Alcohol abuse
* Treatment with glucocorticoids, Glucagon-like peptide-1 (GLP-1) agonists, dipeptidyl peptidase 4 (DPP-4)-inhibitors
* Medical treatment affecting insulin secretion or cardiovascular endpoints
* Liver disease
* Decreased kidney function
* Severe claustrophobia
* Elements incompatible with MR.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2024-05-07 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Coefficient of variation on total blood flow and regional renal perfusion measurements at rest and during isometric muscle exercise, measured by PET/CT with 15-Oxygen labeled water and MRI | Each participant's study day during the span of the study (approximately 5 months)
  No metric unit
Total blood flow at rest and during isometric muscle exercise measured by PET/CT with 15-Oxygen labeled water and MRI | Each participant's study day during the span of the study (approximately 5 months)
  Volume of blood pr unit time, ml/min
Regional renal perfusion at rest and during isometric muscle exercise measured by PET/CT with 15-Oxygen labeled water and MRI | Each participant's study day during the span of the study (approximately 5 months)
  Volume of blood pr unit time pr unit tissue mass, ml/min/g
Regional renal oxygenation at rest and during isometric muscle exercise using MRI | Each participant's study day during the span of the study (approximately 5 months)
  Percentage, fraction
Regional renal extraction of oxygen at rest and during isometric muscle exercise using MRI | Each participant's study day during the span of the study (approximately 5 months)
  Percentage, fraction
Coefficient of variation on regional renal oxygenation and extraction of oxygen measurements at rest and isometric muscle exercise using MRI | Each participant's study day during the span of the study (approximately 5 months)
  No metric unit

CONTACTS AND LOCATIONS:
Overall Officials: Ali Asmar, MD, PhD, Principal Investigator — Bispebjerg Hospital, Department of Clinical Physiology and Nuclear Medicine
Locations (1):
- Bispebjerg Hospital, Department of Clinical Physiology & Nuclear Medicine, Copenhagen, Capital Region, Denmark